CLINICAL TRIAL: NCT01692717
Title: Clinical Assessment Of Association Pharmacokinetics Atorvastatin + Losartana + Hydrochlorothiazide Produced By Lab Hypermarcas S/A In Healthy Subjects
Brief Title: Clinical Assessment Of Association Pharmacokinetics Atorvastatin + Losartana + Hydrochlorothiazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALHHYP0512OR-I; Version 01 May 28, 2012 (Other: LAL Clínica)
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Atorvastatin; hydrochlorothiazide, losartan drug combination; Hydrochlorothiazide; Losartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atorvastatin (Active Comparator): Citalor (Atorvastatin) - Pfizer
  Interventions: Drug: Atorvastatin; Drug: Hydrochlorothiazide + Losartan; Drug: Hydrochlorothiazide + Losartan + Atorvastatin
- Hydrochlorothiazide + Losartan (Active Comparator): Hyzaar (Hydrochlorothiazide + Losartan) - Merck Sharp & Dohme
  Interventions: Drug: Atorvastatin; Drug: Hydrochlorothiazide + Losartan; Drug: Hydrochlorothiazide + Losartan + Atorvastatin
- Atorvastatin + Hydrochlorothiazide + Losartan (Experimental): Polipílula (Atorvastatin + Hydrochlorothiazide + Losartan) - Lab Hypermarcas
  Interventions: Drug: Atorvastatin; Drug: Hydrochlorothiazide + Losartan; Drug: Hydrochlorothiazide + Losartan + Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 10 mg
  Other Names: Citalor
Drug: Hydrochlorothiazide + Losartan — 12.5 mg + 50 mg
  Other Names: Hyzaar
Drug: Hydrochlorothiazide + Losartan + Atorvastatin — 12.5 mg + 50 mg + 10 mg
  Other Names: Polipílula

SUMMARY:
The objective of this clinical study, randomized, crossover is to evaluate the pharmacokinetic profile of the polypill (atorvastatin + lorsatana + hydrochlorothiazide) Laboratory Hypermarcas S / A, in relation to drugs Citalor ® (atovastatina - Pfizer) and Hyzaar ® (losartan + hydrochlorothiazide - Merck Sharp & Dohme) by comparing the serum concentration of analytes unchanged (AT, LS and HCTZ) in healthy subjects.

DETAILED DESCRIPTION:
The pharmacokinetic profile of the drug will also be assessed by comparing the serum concentration of active metabolites following:

* O-hydroxy atorvastatin (2-Hydroxy atorvastatin, O-HAT): metabolite of AT
* carboxylic acid (E-3174, LS-CA): active metabolite of LS

ELIGIBILITY:
Inclusion Criteria:

1. Confirm voluntary participation and agree to all the purposes of the study by signing and dating the IC in two ways;
2. Age between 18 and 55 years, regardless of sex, clinically healthy and present laboratory parameters within normal limits;
3. BMI ≥ 18.5 and ≤ 30.

Exclusion Criteria:

1. Participation in clinical trials in the 12 months preceding the survey;
2. History of hypersensitivity reactions to atorvastatin, losartan hydrochlorothiazide and / or any other ingredients of medicines;
3. Alterations in clinical and laboratory criteria that interfere Principal Investigator on the study results;
4. Presence of pulmonary diseases, cardiovascular, neurological, endocrine, gastrointestinal, genitourinary or other systems;
5. Acute illness during the 07 days preceding the start of the study;
6. Chronic disease that determine drug delivery, such as hypertension, diabetes or any other that requires continuous use of any medicine, including use of vitamins, mineral supplements and OTCs (over-the-counter);
7. Having made regular use of medication in the last 02 weeks before the onset of the study. The use of any medication that does not interfere with the physician's judgment on the pharmacokinetics of the drug under study, will not be considered as an exclusion criterion.
8. Use of medications that interact with any medications association;
9. History of or current use for at least 12 months of tobacco;
10. Current or previous history (under 12 months) of illicit drug use;
11. At the discretion of the Principal Investigator of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
The primary pharmacokinetic parameters for the exercise of comparability will be unchanged dosages of analytes (AT, LS and HCTZ), assessed by AUC, Tmax, Cmax and T1 / 2. | 0h00, 0h15, 0h30, 0h45, 1h00, 1h15, 1h30, 1h45, 2h00, 2h30, 3h00, 3h30, 4h00, 4h30, 5h00, 6h00, 8h00, 10h00, 12h00, 18h00, 24h00, 36h00, 48h00, 56h00 e 72h00.

SECONDARY OUTCOMES:
Pharmacokinetic parameters are side dosages of active metabolites O-HAT and E-3174, measured by AUC, Tmax, Cmax and T1 / 2. | 0h00, 0h15, 0h30, 0h45, 1h00, 1h15, 1h30, 1h45, 2h00, 2h30, 3h00, 3h30, 4h00, 4h30, 5h00, 6h00, 8h00, 10h00, 12h00, 18h00, 24h00, 36h00, 48h00, 56h00 e 72h00.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil